CLINICAL TRIAL: NCT07279077
Title: Node-Sparing Low-Dose Radiotherapy Concurrent With Chemotherapy and PD-1 Inhibitor in pMMR/MSS High-Risk Locally Advanced Colon Cancer: A Prospective, Single-Arm, Phase II Trial
Acronym: MODIFI-L
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sixth Affiliated Hospital, Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Yanxin Luo,MD, MD PHD, Sixth Affiliated Hospital, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025ZSLYEC-669
Record Dates: First submitted 2025-12-01; First posted 2025-12-12 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Colon Cancer; Neoadjuvant Therapies; Immune Checkpoint Therapy; Radiation Therapy
MeSH Terms: conditions — Colonic Neoplasms | interventions — Drug Therapy; Immune Checkpoint Inhibitors

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Node-sparing Low-Dose Radiotherapy Concurrent With Chemotherapy and PD-1 Inhibitor (Experimental): D1, D2: Node-sparing low-dose radiotherapy (1GY*2d) concurrent with chemotherapy (CAPOX) and PD-1 Inhibitor (200mg). 4 cycles, q3w, as total neoadjuvant therapy
  Interventions: Combination Product: Node-Sparing Low-Dose Radiotherapy Concurrent With Chemotherapy and PD-1 Inhibitor

INTERVENTIONS:
Combination Product: Node-Sparing Low-Dose Radiotherapy Concurrent With Chemotherapy and PD-1 Inhibitor — Patients will receive 4 cycles of neoadjuvant therapy: In D1, D2: node-sparing low-dose radiotherapy (1Gy*2d), concurrent with CAPOX chemotherapy and PD-1 inhibitor(200mg). After that, patients will undergo partial colectomy at the site of tumor.

SUMMARY:
Most colorectal cancers belong to the microsatellite stable (MSS) or proficient mismatch repair (pMMR) subtypes, with limited response to PD-1 inhibitors. Radiotherapy can increase the release of tumor-associated antigens, thereby improve responsiveness to PD-1 blockade in MSS/pMMR rectal cancer. Tumor-draining lymph nodes are important sites for PD-1 inhibitors to exert antitumor effects, and studies have reported that direct radiation-induced damage and fibrosis can inhibit lymph node drainage and anti-tumor function. Accumulating evidence indicates that low-dose radiotherapy reprograms the tumor microenvironment (TME), transforming immunosuppressive 'cold' tumors into immunostimulatory 'hot' tumors. This transition is mediated by modulating the gut microbiota, eliciting innate and adaptive immune responses, inhibiting immunosuppressive cells, and promoting the infiltration of T and B lymphocytes.Therefore, this study aims to evaluate whether node-sparing low-dose radiotherapy (1Gy/8f) concurrent with chemotherapy and PD-1 inhibitor can improve the pathological complete response (pCR) rate, enhance tolerability, and improve prognosis in patients with pMMR/MSS high-risk locally advanced colon cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily signed written informed consent.
2. Age ≥ 18 years and ≤ 75 years at the time of enrollment.
3. Eastern Cooperative Oncology Group (ECOG) performance status score of 0 or 1.
4. Life expectancy > 2 years.
5. Histologically confirmed adenocarcinoma of the colon (without squamous or sarcomatoid components).
6. Tumor biopsy immunohistochemistry (IHC) indicates pMMR (proficient Mismatch Repair), defined as positive expression of all four proteins: MSH1, MSH2, MSH6, and PMS2; or genetic testing indicates MSS (Microsatellite Stable).
7. Staged as T4 and/or N+ (Stage IIB-III) according to the AJCC 8th edition, as evaluated by imaging (contrast-enhanced CT or MRI).
8. Prior to enrollment, the subject must be evaluated by a surgeon responsible for the operation based on medical history to confirm eligibility for R0 resection with curative intent.
9. No prior systemic or local anti-tumor therapy for colon cancer before study treatment, including radiotherapy, chemotherapy, immunotherapy, biologics, small molecule targeted therapy, etc.
10. Subjects agree to the collection of tumor tissue and peripheral blood samples required during the screening period and the study process for use in related research.
11. Adequate organ function:

    a) Hematology (no use of blood components or cell growth factors within 7 days prior to the start of study treatment): i. Absolute Neutrophil Count (ANC) ≥ 1.5 × 10⁹/L (1,500/mm³). ii. Platelet count ≥ 100 × 10⁹/L (100,000/mm³). iii. Hemoglobin ≥ 90 g/L. b) Renal: i. Calculated Creatinine Clearance (CrCl) ≥ 50 mL/min (calculated using the Cockcroft-Gault formula: CrCl (mL/min) = {(140 - Age) × Weight (kg) × 0.85 [if female]} / (Serum Creatinine (mg/dL) × 72)).

    ii. Urine protein < 2+ or 24-hour urine protein quantification < 1.0 g. c) Hepatic: i. Serum Total Bilirubin (TBil) ≤ 1.5 × ULN (Upper Limit of Normal). ii. AST and ALT ≤ 2.5 × ULN. iii. Serum Albumin (ALB) ≥ 28 g/L. d) Coagulation: i. International Normalized Ratio (INR) and Activated Partial Thromboplastin Time (APTT) ≤ 1.5 × ULN.

    e) Cardiac Function: i. Left Ventricular Ejection Fraction (LVEF) ≥ 50%.
12. Female subjects of childbearing potential must have a negative urine or serum pregnancy test within 3 days prior to study treatment (if the urine test result cannot confirm negativity, a serum pregnancy test is required, and the serum result prevails). If a female subject of childbearing potential engages in sexual activity with a non-sterilized male partner, she must use an acceptable method of contraception starting from screening and agree to continue using it for 120 days after the last dose of the study drug; cessation of contraception after this point should be discussed with the investigator. Periodic abstinence and rhythm methods are not acceptable forms of contraception.

    1. Women of childbearing potential are defined as women who have not undergone surgical sterilization (i.e., bilateral tubal ligation, bilateral oophorectomy, or hysterectomy) or are not postmenopausal (menopause is defined as at least 12 consecutive months of amenorrhea without an alternative medical cause, with serum Follicle-Stimulating Hormone [FSH] levels within the laboratory reference range for postmenopausal women).
    2. Highly effective contraception refers to methods with a low failure rate (e.g., less than 1% per year) when used consistently and correctly. Not all contraceptive methods are highly effective. In addition to barrier methods, female subjects of childbearing potential must independently use a hormonal contraceptive method (e.g., birth control pills) to ensure pregnancy does not occur.
13. Subjects are willing and able to comply with scheduled visits, treatment plans, laboratory tests, and other study requirements.

Exclusion Criteria:

1. Presence of suspicious metastatic lesions or locally advanced unresectable disease, regardless of disease stage.
2. Subjects who have had other malignancies within 5 years prior to enrollment, excluding colorectal cancer. This excludes subjects with other malignancies cured by local therapy, such as basal or squamous cell skin cancer, superficial bladder cancer, or carcinoma in situ of the breast.
3. Receipt of any investigational drug or investigational device therapy within 4 weeks prior to the first dose of the study drug.
4. Presence of intestinal obstruction, bowel perforation, or intestinal bleeding requiring emergency surgical intervention.
5. Multiple primary colorectal cancers.
6. History of pelvic or abdominal radiotherapy.
7. Inability to swallow pills, malabsorption syndrome, or any condition affecting gastrointestinal absorption.
8. Prior receipt of any systemic or local anti-tumor therapy for locally advanced colon cancer, including radical surgery, chemotherapy, radiotherapy, immunotherapy (including immune checkpoint inhibitors, immune checkpoint agonists, immune cell therapy, or any therapy targeting tumor immune mechanisms), biologics, small molecule targeted therapy, etc.
9. Receipt of non-specific immunomodulatory therapy (e.g., interleukins, interferons, thymosin, tumor necrosis factor, etc., excluding IL-11 used for thrombocytopenia) within 2 weeks prior to study treatment; receipt of traditional Chinese medicine or herbal preparations with anti-tumor indications within 1 week prior to study treatment.
10. Active autoimmune disease requiring systemic treatment (e.g., disease-modifying antirheumatic drugs, corticosteroids, immunosuppressants) within the past two years. Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement for adrenal or pituitary insufficiency) is not considered systemic treatment.
11. History of non-infectious pneumonitis or pneumonia requiring systemic glucocorticoid treatment, or current history of interstitial lung disease.
12. History of severe bleeding tendency or coagulation disorders; patients requiring prior or current long-term anticoagulation therapy (e.g., atrial fibrillation patients meeting CHADS2 score ≥ 2).
13. Current uncontrolled comorbidities, including but not limited to decompensated liver cirrhosis, nephrotic syndrome, uncontrolled metabolic disorders, severe active peptic ulcer disease or gastritis, or psychiatric/social conditions that would limit the subject's compliance with study requirements or affect their ability to provide written informed consent.
14. History of myocarditis, cardiomyopathy, or malignant arrhythmia.

    1. Within 12 months prior to study treatment: unstable angina requiring hospitalization, congestive heart failure, or vascular disease (e.g., aortic aneurysm requiring surgical repair or peripheral venous thrombosis), or other cardiac damage that may affect the safety evaluation of the study drug (e.g., poorly controlled arrhythmia, myocardial infarction, or ischemia).
    2. Within 6 months prior to study treatment: history of esophageal/gastric varices, severe ulcer, unhealed wound, gastrointestinal perforation, abdominal fistula, gastrointestinal obstruction, intra-abdominal abscess, or acute gastrointestinal bleeding.
    3. Within 6 months prior to study treatment: any arterial thromboembolic event, NCI CTCAE v5.0 Grade 3 or higher venous thromboembolism, transient ischemic attack (TIA), cerebrovascular accident (stroke), hypertensive crisis, or hypertensive encephalopathy.
    4. Within 1 month prior to study treatment: acute exacerbation of chronic obstructive pulmonary disease (COPD).
    5. Current hypertension with systolic BP ≥ 160 mmHg or diastolic BP ≥ 100 mmHg despite oral antihypertensive medication.
15. Active or documented history of inflammatory bowel disease (e.g., Crohn's disease, ulcerative colitis, or chronic diarrhea).
16. Severe infection within 4 weeks prior to study treatment, including but not limited to comorbidities requiring hospitalization, sepsis, or severe pneumonia; active infection requiring systemic anti-infective treatment within 10 days prior to study treatment (excluding antiviral treatment for Hepatitis B or C).
17. Major surgery or severe trauma within 30 days prior to study treatment; minor local surgery within 3 days prior to study treatment (excluding Peripherally Inserted Central Catheter [PICC] or Central Venous Catheter [CVC] placement).
18. History of immunodeficiency; positive HIV antibody test; currently receiving long-term systemic corticosteroids or other immunosuppressants.
19. Known active tuberculosis (TB); subjects suspected of having active TB must undergo clinical examination to exclude it (e.g., sputum smear, chest X-ray); known active syphilis infection.
20. Known history of allogeneic organ transplantation or allogeneic hematopoietic stem cell transplantation.
21. Untreated active Hepatitis B subjects (HBsAg positive and HBV-DNA > 1000 copies/mL [200 IU/mL] or above the lower limit of detection); subjects with Hepatitis B are required to receive anti-HBV treatment during the study treatment period. Active Hepatitis C subjects (HCV antibody positive and HCV-RNA levels above the lower limit of detection).
22. Receipt of live vaccines within 30 days prior to study treatment, or planned receipt of live vaccines during the study period.
23. Known allergy to any component of the study drugs; known history of severe hypersensitivity reactions to other monoclonal antibodies.
24. Known history of psychiatric illness, drug abuse, alcohol abuse, or substance abuse.
25. Pregnant or lactating women.
26. Prior or current presence of any disease, treatment, or laboratory abnormality that may confound study results, affect the subject's full participation in the study, or where participation is not in the subject's best interest.
27. Local or systemic diseases not caused by malignancy; or diseases/symptoms secondary to the tumor that lead to high medical risk and/or uncertainty in survival evaluation, such as tumor-related leukemoid reaction (WBC > 20 × 10⁹/L), manifestations of cachexia (e.g., known weight loss of > 10% in the 3 months prior to screening), BMI ≤ 18 (BMI = Weight [kg] / Height [m²]), etc.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2025-11-26 (Actual); Primary Completion 2030-11-25 (Estimated); Study Completion 2031-12-30 (Estimated)

PRIMARY OUTCOMES:
Pathological Complete Response(pCR) Rate | From enrollment to 2-4 weeks after surgery
  Evaluate whether 8Gy/8F node-sparing low-dose radiotherapy concurrent with chemotherapy and PD-1 inhibitor as total neoadjuvant therapy can better improve the pathological complete response(pCR) rate or not in colon cancer.

SECONDARY OUTCOMES:
Tumor regression grade (TRG) | From enrollment to 2-4 weeks after surgery
Tumor downstaging rate | From enrollment to 2-4 weeks after finishing preoperative treatment
R0 resection rate | From enrollment to 2-4 weeks of surgery
3-year overall survival (OS) rate | From enrollment to 3 years after finishing Surgery
Event-Free Survival (EFS) | From enrollment to 3 years after finishing Surgery
3-year distant metastasis rate | From enrollment to 3 years after finishing Surgery
3-year local recurrence rate | From enrollment to 3 years after finishing Surgery

CONTACTS AND LOCATIONS:
Locations (1):
- The Sixth Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No